CLINICAL TRIAL: NCT05412394
Title: Phase-2 Trial of 5mg/kg/Week Prednisolone in Young Boys With DMD
Brief Title: Once Weekly Infant Corticosteroid Trial for DMD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anne M. Connolly (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Muscular Dystrophy Association (Other); University of Texas (Other); Virginia Commonwealth University (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor-Investigator, Anne M. Connolly, Chief of Division of Neurology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Infant Steroid Phase II
Record Dates: First submitted 2022-02-02; First posted 2022-06-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Steroid; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): This is a one-arm study and the group of subjects are all experimental and will receive drug.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Liquid, 5mg/kg per week, for one year
  Other Names: Corticosteroid

SUMMARY:
The hypothesis tested here is that a lower dose of intermittent oral corticosteroids (5mg/kg/week) will be equally effective to the 10mg/kg/week dose.

DETAILED DESCRIPTION:
The investigators know that the muscle destruction from Duchenne muscular dystrophy (DMD) begins in infancy and we previously demonstrated that motor decline in infancy compared to typically developing infants reflects that destruction. Because of the known side effects of daily corticosteroids, most physicians do not begin treatment until age 3-5 years. Most side effects (Cushingoid faces, linear growth arrest, and bone density loss) did not happen in infants and in ambulatory boys in two separate studies. However, in infants and young boys taking (10mg/kg/week), 56% of infants and young boys did have an increase in weight percentile compared to baseline. This study will test this lower dose of prednisolone (5mg/kg/week) in an unblinded study in infants and young DMD boys (ages 1 through 30 months) to determine if equal efficacy can be achieved with fewer side effects. The primary outcome for this study will be gross motor function. The study team will enroll boys from age 1 month through 30 months and follow each for two years. We will assess gross motor function using three outcome measures: the Bayley-4 Scales of Infant and Toddler Development (Bayley-4) and the newly developed Neuromuscular Gross Motor Outcomes (GRO) and the NorthStar Ambulatory Assessment (NSAA). The one-year outcome will be the change in the Bayley-4 Scaled Score and the two-year outcome will be the change in the GRO score. This study will determine if a lower dose is equally effective and if that dose may lessen the weight gain seen in about half of the infants in the first study. Both the Bayley-4 and the GRO allow assessment of gross motor function and are feasible in all boys with DMD under the age of 42 months. In addition, the GRO allows continued assessment of motor function across a wide age span which will allow this cohort to be followed for two full years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 1 month through 30 months
* Weakness consistent with Duchenne on exam, creatine kinase ≥ 20 times the upper limit of normal, and genetic mutation known to be causative for DMD.

Exclusion Criteria:

* Prior treatment with Glucocorticosteroids

Ages: 1 Month to 30 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The change from baseline to 24 months for the Gross Motor Scaled Score. | Baseline visit to 24 month visit
  Neuromuscular Gross Motor Outcome (GRO): The Neuromuscular GRO is a gross motor outcome measure developed to assess whole body strength, motor development, and function for all levels of ability across the lifespan in those diagnosed with neuromuscular disease. Items are administered following the developmental sequence, as appropriate for age and ability. Maximum score is 100 points.

SECONDARY OUTCOMES:
Language (expressive and receptive), Social and Fine Motor skills at 24 months as assessed by the Bayley-4 Scales of Infant and Toddler Development | Baseline visit to 24 month visit
  The Bayley Scales of Infant and Toddler Development (Bayley-4) are recognized internationally as a comprehensive tool to assess children from as young as 15 days old. With Bayley-4, it is possible to obtain detailed information from non-verbal children as to their functioning. Children are assessed in the five key developmental domains of cognition, language (receptive and expressive), & motor (fine and gross).
Linear growth | Baseline visit to 24 month visit
  We have previously shown that all infants and young children treated with 10mg/kg/week did maintain their linear growth. This protocol is designed to determine also if the lower dose will still maintain benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Connolly, MD, Principal Investigator — Nationwide Children's Hospital
Locations (4):
- United States (4):
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas Southwestern, Dallas, Texas